CLINICAL TRIAL: NCT03785067
Title: Triple Therapy Prevention of Recurrent Intracerebral Disease EveNts Trial (TRIDENT) Cognitive Sub-Study
Acronym: TRIDENT COG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Contractual and financial issues.
Sponsor: The George Institute (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: TRIDENT COG
Record Dates: First submitted 2018-12-06; First posted 2018-12-24 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Decline; Intracerebral Hemorrhage; Dementia, Vascular; Cerebral Small Vessel Diseases; Hypertension; Stroke Hemorrhagic
Keywords: TRIDENT
MeSH Terms: conditions — Cognitive Dysfunction; Cerebral Hemorrhage; Dementia, Vascular; Cerebral Small Vessel Diseases; Hypertension; Hemorrhagic Stroke | interventions — Telmisartan; Amlodipine; Indapamide

STUDY DESIGN:
Intervention Model Description: Main Study: Multicentre, international, double-blinded, placebo-controlled, parallel-group, randomised controlled trial.
  Sub-Study: Multicentre, international, single-arm trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Main Study: Participants are double-blinded. Sub-Study: No blinding to neuropsychological assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple Pill (Active Treatment) (Experimental): Main Study: Fixed low-dose combination BP-lowering pill ("Triple Pill") telmisartan 20mg + amlodipine 2.5mg + indapamide 1.25mg
  Sub-Study: single-arm
  Interventions: Drug: telmisartan 20mg + amlodipine 2.5mg +indapamide 1.25mg
- Placebo (Placebo Comparator): Main Study: Matched placebo, received via blinded study capsules
  Sub-Study: single-arm
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: telmisartan 20mg + amlodipine 2.5mg +indapamide 1.25mg — 1 capsule taken orally once daily for 36 months
  Other Names: Triple Pill
  Arms: Triple Pill (Active Treatment)
Drug: Placebo oral capsule — 1 capsule taken orally once daily for 36 months
  Arms: Placebo

SUMMARY:
A Sub-Study of an investigator initiated and conducted, multicentre, international, double-blinded, placebo-controlled, parallel-group, randomised controlled trial (TRIDENT) to determine the effect of more intensive long-term blood pressure control, provided by a fixed low-dose combination blood pressure lowering pill ("Triple Pill") strategy on top of standard of care, for slowing memory decline as measured by Cambridge Neuropsychological Test Automated Battery (CANTAB), in patients with a history of acute stroke due to intracerebral haemorrhage (ICH).

DETAILED DESCRIPTION:
Cognitive decline and dementia in ICH is high due to the common underlying vasculopathy of cerebral small vessel disease (CSVD). However, in general, detailed cognitive outcomes in ICH have been neglected, possibly due to the high mortality rate of ICH (up to 60% within the first year).

Blood pressure (BP) management in those with ICH has been suboptimal. Most hypertensive patients need more than two medications. Combination therapy may improve adherence and BP reduction and reduce cardiovascular (CV) event rates. In the main TRIDENT study, it is hypothesised that a fixed low-dose triple combination BP-lowering agent, termed the 'Triple Pill' will prevent recurrent stroke. The Triple Pill is composed of a single capsule containing either a combination of telmisartan 20 mg, amlodipine 2.5 mg and indapamide 1.25 mg, or placebo.

In addition to achieving optimal BP control, the Triple Pill also has the capacity to slow cognitive decline and dementia in ICH survivors. Research shows that elevated BP is associated with Alzheimer's disease and vascular dementia, even after accounting for prior stroke or transient ischaemic attack, and large scale prospective studies have shown a 50% reduction in dementia when BP is managed appropriately

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for, randomised and continuing in the TRIDENT Main Study
2. Must be able to attend the site conducting the cognitive assessments. In Sydney, this will either be at the same site as where TRIDENT study is conducted or at the BMC, University of Sydney, Camperdown.
3. Ability and willingness to undergo neuropsychological testing (i.e. have no major visual, auditory or motor impairments)
4. Language spoken compatible with CANTAB administration (i.e. CANTAB will be administered in the local language(s) of the country in question. E.g. in Australia, the CANTAB will only be administered in English).
5. Provision of written informed consent

Exclusion Criteria:

1. Study medication has been permanently stopped prior to or at the 6-month visit of the TRIDENT main study
2. Informant Questionnaire for Cognitive Decline in the Elderly (IQCODE) score of 3.313 or higher
3. Cognitive performance indicative of dementia at 6-month TRIDENT main study visit defined by Montreal Cognitive Assessment (MoCA) score less than 2414.
4. Evidence of rapid deterioration suggestive of dementia by decline of 3 points in MoCA assessments between randomisation and the 6-month study visit in the TRIDENT main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Memory as measured by the Cambridge Neuropsychological Test Automated Battery (CANTAB) Paired Associates Learning (PAL) subtest | Baseline, 18 and 36 months
  Raw scores and z-scores will be used. Change scores on the CANTAB PAL will be computed between baseline, 18 and 36 months (primary endpoint).

SECONDARY OUTCOMES:
Change scores will be computed for CANTAB Rapid Visual Information Processing (RVP) | Baseline, 18 and 36 months
  Change scores will be computed for CANTAB RVP between baseline, 18 and 36 months
Change scores will be computed for CANTAB Multi-tasking Test (MTT) | Baseline, 18 and 36 months
  Change scores will be computed for CANTAB MTT between baseline, 18 and 36 months
Change scores will be computed for gold-standard neuropsychological assessments | Baseline, 18 and 36 months
  Change scores will be computed for gold-standard neuropsychological assessment between baseline, 18 and 36 months
Diagnosis of all-cause dementia | 36 months
  Diagnosis of all-cause dementia as determined by consensus of three blinded adjudicators based on established criteria following collection of data of the 3-year study period

CONTACTS AND LOCATIONS:
Overall Officials: Prof Craig Anderson, Principal Investigator — The George Institute; Prof Sharon Naismith, Principal Investigator — University of Sydney
Locations (4):
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal Melbourne Hospital, Melbourne, Victoria
- Radboud University Medical Center, Nijmegen, Netherlands